CLINICAL TRIAL: NCT07124975
Title: Impact of Comparing Treatment Status With Other Patients on Treatment Adherence in CPAP Therapy.
Brief Title: Impact of Comparing Treatment Status With Other CPAP Users
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kimihiko Murase (Other)
Responsible Party: Sponsor-Investigator, Kimihiko Murase, Assistant Professor, Kyoto University Hospital
Organization: Kyoto University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C1736
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Sleep Apnea; Obstructive Sleep Apnea
Keywords: CPAP adherence
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine treatment data feedback group (Active Comparator): In this group, feedback will be provided to participants by mail on monthly basis, including the proportion of days with CPAP usage ≥4 hours per day and the average daily CPAP usage time.
  Interventions: Behavioral: CPAP data feedback
- Treatment data comparison group (Experimental): In this group, feedback will be provided as in the routine treatment data feedback group. In addition to this information, aggregated results for all participants (proportion of days with CPAP usage ≥4 hours per day and average daily usage time) and the participant's ranking based on these aggregated data will also be provided as feedback.
  Interventions: Behavioral: Comparison of the treatment data with other patients; Behavioral: CPAP data feedback

INTERVENTIONS:
Behavioral: Comparison of the treatment data with other patients — In this group, feedback will be provided as in the routine treatment data feedback group. In addition to this information, aggregated results for all participants (proportion of days with CPAP usage ≥4 hours per day and average daily usage time) and the participant's ranking based on these aggregated data will also be provided as feedback.
  Arms: Treatment data comparison group
Behavioral: CPAP data feedback — Participants will receive monthly feedback on their CPAP therapy treatment data (usage time and the proportion of days with >4 hours of use) via mail or email for 6 months.

SUMMARY:
The objective of this study is to evaluate whether comparing a patient's own CPAP usage data with that of other patients improves CPAP adherence in patients who have been undergoing long-term CPAP therapy for sleep apnea. Eligible participants are patients who have been on CPAP therapy with remote monitoring of treatment data enabled for at least three months. Participants will be randomly assigned to one of two groups: (1) routine treatment data feedback group, or (2) treatment data comparison group. In both groups, feedback will be provided to participants by mail on monthly basis, including the proportion of days with CPAP usage ≥4 hours per day and the average daily CPAP usage time. In the treatment data comparison group, in addition to this information, aggregated results for all participants (proportion of days with CPAP usage ≥4 hours per day and average daily usage time) and the participant's ranking based on these aggregated data will also be provided as feedback. The observation period will be six months after initiation of the intervention, and changes in treatment adherence before and after the intervention will be assessed.

ELIGIBILITY:
Eligibility criteria:

* The patient has been diagnosed with SAS and has initiated CPAP therapy according to the criteria of Japanese public health insurance system(i.e., Apnea hypopnea index (AHI) >= 20/h by polysomnography, or respiratory event index (REI) is >= 40/h by portable monitoring device at the time of OSA diagnosis).
* The patient makes regular outpatient visits for the continuation of CPAP therapy according to the requirements for the coverage of Japanese public health insurance.
* At least three months have passed since the introduction of a CPAP remote monitoring system, and the researchers can confirm CPAP adherence online.
* The patient has mailing address necessary for sending feedback by post or email.

Exclusion Criteria:

* Treatment adherence is already sufficiently good, with little need for further improvement. (Defined as a proportion of days with >4 hours of CPAP use of 90% or higher, and an average daily usage time >=7 hours over the past month.)
* No CPAP usage at all during the past month (for example, due to business trips, caring for family members, or other social reasons resulting in an inability to use CPAP, and for whom improvement in adherence through this intervention is not expected).
* Working night shifts twice or more a week.
* Patients with cognitive impairment

Intervention Details

1. When a patient who is a potential participant visits the outpatient clinic for continued CPAP therapy, their CPAP adherence during the previous month will be checked.
2. If the patient's background and CPAP adherence over the previous month meet the inclusion criteria, informed consent will be obtained from the patient.
3. After the number of patients who have provided consent reaches the planned sample size, a postal item will be sent to confirm the accuracy of the participant's address. The mailing will include a postcard for reply or QR code that allows the research team to verify that the participant has received the item. Participants whose receipt of the mailing can be confirmed will be eligible for randomization.
4. Participants will be randomly assigned to either the control group (receiving only information about their own CPAP adherence) or the peer comparison group (receiving information about their own adherence plus the summary of adherence data from all participants).
5. Thereafter, for six months, participants will receive by mail monthly information about their CPAP adherence. Each mailing will include a postcard for reply and a QR code that allow participants to notify the researchers that they have opened the mailing.

In the control group, the following information will be provided:(1) Average daily CPAP usage time in the previous month, and (2) Percentage of days with CPAP usage more than or equal to 4 hours per day.In the peer comparison group, in addition to the above, the following information will be provided: (3) Mean daily CPAP usage time among all participants, (4) Percentage of days with CPAP usage ≥ 4 hours per day among all participants, and (5) Participant's rank among all participants based on average daily CPAP usage time.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improvement in CPAP adherence | 6 months from the start of the interventions
  CPAP adherence during the six months following initiation of the intervention will be compared with adherence during the three months before obtaining consent. Improvement in adherence will be defined as meeting either of the following criteria: (1) an increase of ≥10% in the proportion of days with ≥4 hours of CPAP use, or (2) an increase of ≥40 minutes in the average daily usage time.

SECONDARY OUTCOMES:
CPAP adherence | 6 months
  Change in the proportion of days with >=4 hours of CPAP use
CPAP adherence | 6 months
  Change in the average daily usage time
daytime sleepiness | 6 months
  Daytime sleepiness will be assessed using a questionnaire at the start and end of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: Undecided
Due to ethical considerations, the study data will be available upon request by contacting the corresponding author. The corresponding author will verify whether the request is subject to confidentiality obligations.